CLINICAL TRIAL: NCT06639672
Title: Neoadjuvant Chemotherapy Combined With PD-1 Inhibitor and Different Radiotherapy Fractionations for HR+/HER2- Breast Cancer: A Phase II Study
Brief Title: Neoadjuvant Chemotherapy + PD-1 Inhibitor+Different Radiotherapy Fractionations for HR+/HER2- Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Liu (Other)
Responsible Party: Sponsor-Investigator, Lei Liu, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20241777
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: HR+HER2- Breast Cancer
Keywords: HR+/HER2- breast cancer; Neoadjuvant chemotherapy; Immunotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): 8Gy x 3f + Chemotherapy+Immunotherapy
  Interventions: Drug: Chemotherapy+PD-1 inhibitor+8Gy x 3f
- Arm 2 (Experimental): 16Gy x 1f + Chemotherapy+Immunotherapy
  Interventions: Drug: Chemotherapy+PD-1 inhibitor+16Gy x 1f
- Arm 3 (Experimental): 2.76Gy x 15f + Chemotherapy+Immunotherapy
  Interventions: Drug: Chemotherapy+PD-1 inhibitor+2.67Gy x 15f
- Arm 4 (Experimental): 0.5Gy x 12-18f + Chemotherapy+Immunotherapy
  Interventions: Drug: Chemotherapy+PD-1 inhibitor+0.5Gy x 12-18f

INTERVENTIONS:
Drug: Chemotherapy+PD-1 inhibitor+8Gy x 3f — Radiotherapy: 8Gy x 3f, once every other day; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle. Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: Arm 1
Drug: Chemotherapy+PD-1 inhibitor+16Gy x 1f — Radiotherapy: 16Gy x 1f; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle. Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: Arm 2
Drug: Chemotherapy+PD-1 inhibitor+2.67Gy x 15f — Radiotherapy: 2.67Gy x 15f; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle. Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: Arm 3
Drug: Chemotherapy+PD-1 inhibitor+0.5Gy x 12-18f — Radiotherapy: 0.5Gy x 12-18f; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle. Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: Arm 4

SUMMARY:
For the hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-) subtype of breast cancer, although surgical, radiotherapy, and endocrine treatments have shown better survival, this subtype has a relatively poor response to neoadjuvant chemotherapy and immunotherapy, with an approximately pCR of 20%. The low immunogenicity result in suboptimal pCR and objective response rates for this group. Therefore, there is an urgent need to explore new, highly effective, and low-toxicity treatment strategies to further improve the efficacy of HR+/HER2- breast cancer. Radiotherapy has systemic immune regulatory effects by promoting the release of antigens from tumor cells, enhancing T-cell infiltration, and directly killing tumor cells. Therefore, this study aims to investigate the efficacy and safety of chemotherapy combined with PD-1 inhibitor and different radiotherapy fractionations in the neoadjuvant treatment of HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed HR+/HER2- breast cancer
* 2. cT1c-2N1-2M0 or cT3N0-2M0（AJCC 7th）
* 3. ECOG performance status of 0-1;
* 4. Adequate bone marrow function, defined as: Hb ≥ 9.0 g/dL (90 g/L); ANC ≥ 1,500/mcL (1.5 × 10^9/L); PLT ≥ 100,000/mcL (100 × 10^9/L) and no blood transfusion within 3 weeks or growth factor (G-CSF, EPO) therapy within 2 weeks prior to dosing;
* 5. Adequate liver function, defined as: TBIL ≤ 1.5× upper limit of normal (ULN); If no liver metastases, AST and ALT ≤ 2.5× ULN; if liver metastases are present, AST or ALT ≤ 3.0× ULN; ALP ≤ 1.5× ULN; if liver metastases ≤ 2× ULN; Serum albumin ≥ 30g/L;
* 6. Adequate coagulation function: INR or PT, APTT ≤ 1.5× ULN. Participants on anticoagulant therapy should have these laboratory indices closely monitored;
* 7. Adequate renal function, defined as creatinine ≤ 1.5× ULN or Ccr ≥ 50 mL/min calculated using the Cockcroft-Gault formula corrected for body surface area;
* 8. Baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO);
* 9. No severe organic heart disease or arrhythmias;
* 10. Women of childbearing potential (aged 15-49 years) must have a negative pregnancy test within 7 days before starting treatment. Both male and female participants of reproductive potential must agree to use effective contraceptive measures during the study period and for 3 months after discontinuation of treatment;
* 11. Voluntary signed informed consent by the study participant.

Exclusion Criteria:

* 1. Patients with a history of mental illness or those diagnosed with mental disorders at the time of enrollment in the clinical trial.
* 2. Patients with communication barriers due to confusion, aphasia, intellectual disability, or other reasons that prevent them from responding normally.
* 3. Poorly controlled tumor-related pain.
* 4. Patients participating in other clinical studies simultaneously.
* 5. Patients with active or past autoimmune diseases or immunodeficiencies, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* 6. A history of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on chest CT scans at screening.
* 7. Active pulmonary tuberculosis.
* 8. Severe cardiovascular diseases occurring within 3 months prior to the start of study treatment (e.g., NYHA class II or higher heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmias, or unstable angina.
* 9. Patients who underwent significant surgical procedures, other than diagnostic surgeries, within 4 weeks prior to the start of the study treatment, or are expected to require significant surgical procedures during the study period.
* 10. Patients who had malignant tumors other than breast cancer within the last 5 years, except for malignancies in the study that have negligible risks of metastasis or death , such as adequately treated cervical carcinoma in situ, non-melanoma skin cancer, ductal carcinoma in situ, or stage I uterine cancer.
* 11. Patients who experienced severe infections within 4 weeks prior to the start of the study treatment, including but not limited to those requiring hospitalization due to infections, bacteremia, severe pneumonia, or any active infection that may impact patient safety.
* 12. Patients who have previously received allogeneic stem cell or solid organ transplants.
* 13. Any other diseases, metabolic dysfunctions, physical examination abnormalities, or clinical laboratory abnormalities that contraindicate the use of the study drug, may affect the interpretation of results, or pose a high risk of treatment complications for the patient.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
pCR | Up to approximately 2 years
  The percentage of patients showing no evidence of invasive cancer cells in the tissue samples after treatment

SECONDARY OUTCOMES:
Ipsilateral breast recurrence or local regional recurrence | 5 year
  The percentage of patients experiencing a recurrence of cancer in the same breast or in the nearby lymph nodes
Overall survival | 5 year
  The time from the start of treatment until the occurrence of death
Distant metastasis-free survival | 5 year
  the time from the start of treatment until the occurrence of distant metastasis
Incidence of Treatment-Emergent Adverse Events | Up to approximately 1 years
  the incidence of adverse events

IPD SHARING:
Plan to Share IPD: No